CLINICAL TRIAL: NCT02550119
Title: A Pilot Study to Evaluate the Safety and Efficacy of Aprepitant in Combination With Dolasetron and Dexamethasone for the Prevention of Nausea and Vomiting Following Oxaliplatin-containing Regimen Which Includes 5-FU.
Brief Title: Dolasetron Mesylate and Dexamethasone With or Without Aprepitant in Preventing Nausea and Vomiting in Patients Undergoing Oxaliplatin-Containing Chemotherapy for Gastrointestinal Malignancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3C-06-1; NCI-2012-01740 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-06-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-09-13; First posted 2015-09-15 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Malignant Digestive System Neoplasm; Nausea and Vomiting
MeSH Terms: conditions — Gastrointestinal Neoplasms; Nausea; Vomiting | interventions — Aprepitant; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; dolasetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (aprepitant, dolasetron mesylate, dexamethasone) (Experimental): Patients receive dolasetron mesylate PO or IV, dexamethasone PO or IV, and aprepitant PO 1 day before chemotherapy and dexamethasone PO and aprepitant PO on days 2 and 3 after chemotherapy begins during course 2-3.
  Interventions: Drug: Aprepitant; Drug: Dexamethasone; Drug: Dolasetron Mesylate
- Arm II (placebo, dolasetron mesylate, dexamethasone) (Placebo Comparator): Patients receive dolasetron mesylate and dexamethasone as in Arm I and placebo PO 1 day before chemotherapy and dexamethasone PO and placebo PO on days 2 and 3 after chemotherapy begins during courses 2-3.
  Interventions: Drug: Dexamethasone; Drug: Dolasetron Mesylate; Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant — Given PO
  Other Names: Emend; L-754030; MK-0869; ONO-7436
  Arms: Arm I (aprepitant, dolasetron mesylate, dexamethasone)
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Dolasetron Mesylate — Given PO or IV
  Other Names: Anzemet; MDL 73,147EF
Drug: Placebo — Given PO
  Other Names: PLCB; sham therapy
  Arms: Arm II (placebo, dolasetron mesylate, dexamethasone)

SUMMARY:
This randomized pilot clinical trial dolasetron mesylate and dexamethasone with or without aprepitant in preventing nausea and vomiting in patients undergoing oxaliplatin-containing chemotherapy for gastrointestinal malignancy. Antiemetic drugs may help lessen or prevent nausea and vomiting in patients treated with chemotherapy. It is not yet known whether giving aprepitant together with dolasetron mesylate and dexamethasone is more effective than dolasetron mesylate and dexamethasone alone in preventing nausea and vomiting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the incidence and severity of acute and delayed nausea and vomiting associated with oxaliplatin-containing regimens in patients with gastrointestinal (GI) malignancy.

II. To estimate the percent of patients who have experienced nausea and vomiting with their first or second cycle of oxaliplatin-containing regimen, and would consent to randomization to standard antiemetic therapy with or without aprepitant.

III. To obtain preliminary data on the safety and efficacy of aprepitant, in combination with dolasetron (dolasetron mesylate) and dexamethasone, in patients receiving oxaliplatin-containing regimen.

IV. To report on medication compliance with antiemetic medications (dexamethasone and aprepitant or placebo) scheduled to be taken at home on days 2 and 3 for all randomized patients (day 1 = day of treatment).

OUTLINE: Patients receive standard antiemetics comprising dolasetron mesylate orally (PO) or intravenously (IV) and dexamethasone PO or IV during course 1 of oxaliplatin-containing chemotherapy. Patients experiencing any grade 1-4 nausea and vomiting* are randomized to 1 of 2 treatment arms.

ARM I: Patients receive dolasetron mesylate PO or IV, dexamethasone PO or IV, and aprepitant PO 1 day before chemotherapy and dexamethasone PO and aprepitant PO on days 2 and 3 after chemotherapy begins during course 2-3.

ARM II: Patients receive dolasetron mesylate and dexamethasone as in Arm I and placebo PO 1 day before chemotherapy and dexamethasone PO and placebo PO on days 2 and 3 after chemotherapy begins during courses 2-3.

In both arms, treatment continues in the absence of unacceptable toxicity.

NOTE: * Patients not developing nausea and vomiting until the second course of treatment are also randomized during courses 3 and 4 of chemotherapy.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis of GI malignancy and who are scheduled to receive their initial treatment with an oxaliplatin-containing regimen in combination with 5-fluorouracil; these include combinations such as fluorouracil, oxaliplatin, and leucovorin calcium (FOLFOX), FOLFOX + bevacizumab, FOLFOX + cetuximab
* Standard antiemetic therapy with initial treatment must include the dolasetron and dexamethasone; the minimum adequate doses include either:

  * Dolasetron (Anzemet) 100mg PO/IV or 1.8mg/kg IV AND
  * Dexamethasone (Decadron) 10mg PO/IV
* Patient must agree, as part of the informed consent, to keep a journal of the episodes of nausea, vomiting, retching, and amount of rescue medications used on days 1 to 5 (day 1 = day of treatment)
* Signed informed consent

Exclusion Criteria:

* Allergy or intolerance to dolasetron and dexamethasone
* Use of another antiemetic agent (5HT3 antagonists, phenothiazines, butyrophenones, cannabinoids, metoclopramide, or corticosteroids) within 72 hours of day 1 of the study
* An episode of vomiting or retching within 24 hours before the start of the initial treatment with oxaliplatin-containing regimen
* Severe concurrent illness other than neoplasia
* Gastrointestinal obstruction or an active peptic ulcer
* Radiation therapy to the abdomen or pelvis within 1 week before or after day 1 of the study
* Absolute neutrophil count of less than 1.5 x 10^9/L (unless physician approves to proceed with chemotherapy) or
* Platelets less than 100 x 109/L (unless physician approves to proceed with chemotherapy)
* Total bilirubin > 2 x upper limits of normal
* Patients who are pregnant or breast feeding
* Patients who are non-English speaking
* Patients with cancer-induced nausea and vomiting grade 1 or greater using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-04-19 (Actual); Primary Completion 2010-04-01 (Actual); Study Completion 2010-04-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete response, defined as no emesis and no use of rescue medication | Within the first 24 hours of treatment (day 1)
  We will summarize the incidence, severity and time of onset of all nausea and vomiting experienced by all patients who received any oxaliplatin. The complete response rates in both arms will be calculated with 95% confidence intervals.

SECONDARY OUTCOMES:
Proportion of patients who agreed to be randomized out of all patients who qualify for randomization | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Betty Chan, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States